CLINICAL TRIAL: NCT02533310
Title: Single-session Gamified Virtual Reality Exposure Therapy for Spider Phobia vs. Traditional Exposure Therapy: a Randomized Controlled Non-inferiority Trial
Brief Title: Virtual Reality Immersive Method for Spider (Phobia) Exposure Therapy (VIMSE)
Acronym: VIMSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Responsible Party: Principal Investigator, Per Carlbring, Professor of Psychology and Head of subdivision of Clinical Psychology, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIMSE
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Phobia, Specific
Keywords: Specific phobia; Exposure therapy; Virtual reality; Randomized controlled trial
MeSH Terms: conditions — Phobia, Specific

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OST treatment with in-vivo spiders (Experimental): OST consists of increasingly intense interactions with an in-vivo phobic stimuli and human therapist non-phobic behavior modelling.
  Interventions: Other: OST treatment with in-vivo spiders
- VR-OST treatment with virtual spiders (Experimental): VR-OST consists of simulated OST treatment without the use of live spiders and with the support of a virtual therapist.
  Interventions: Other: VR-OST treatment with virtual spiders

INTERVENTIONS:
Other: OST treatment with in-vivo spiders — Subjects are exposed to phobic stimuli with the aid of a trained psychotherapist during a session of maximum 3 hrs duration. The intensity of exposure is increased in four sequential steps, 1. learning to catch a spider with a glass and paper, 2. touching a spider, 3. letting a spider walk on your hand, 4. letting a spider walk on your body. These stages repeat with increasingly larger spiders. The goal of therapy is not absolute symptom reduction but sufficient reduction to allow the individual to expose themselves in everyday situations.
  Arms: OST treatment with in-vivo spiders
Other: VR-OST treatment with virtual spiders — The VR-OST treatment introduces a virtual gamified version of OST treatment using a modern virtual reality headset. Individuals advance themselves through increasing levels of exposure intensity with the assistance of an automated virtual therapist.
  Arms: VR-OST treatment with virtual spiders

SUMMARY:
The aim of this study is to examine the efficacy of virtual reality exposure therapy as a treatment for specific phobia (spiders). A gamified virtual reality simulation of one-session therapy (VR-OST) will be compared to the gold-standard treatment in the form of traditional one-session phobia treatment (OST) using in-vivo stimuli. This study was powered to detect a non-inferiority margin of a 2-point difference between groups.

ELIGIBILITY:
Inclusion Criteria:

* Score of 10 or less in Behavioral Approach Test
* Individual meeting DSM-5 criteria according to interview for primary diagnosis of specific phobia, spider
* Swedish residency
* Fluent in Swedish

Exclusion Criteria:

* Ongoing psychotherapy
* Ongoing psychotropic medication (unless stabilized for three months)
* Indication of suicidal ideation, as assessed by item 9 of the PHQ-9
* Meets criteria for alcohol or substance use disorder
* Meets criteria for serious mental disorder, such as bipolar disorder, schizophrenia or psychosis
* Balance and/or eyesight problems (such as lack of stereoscopic vision) that could interfere with VR treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Behavioral Approach Test (BAT) | Change from baseline on BAT (1 week)
  The BAT consists of 13 approach steps measuring intensity of phobia symptoms, from approaching a few metres from to holding a spider.
Behavioral Approach Test (BAT) | Change from baseline on BAT (12 week)
  The BAT consists of 13 approach steps measuring intensity of phobia symptoms, from approaching a few metres from to holding a spider.
Behavioral Approach Test (BAT) | Change from baseline on BAT (52 week)
  The BAT consists of 13 approach steps measuring intensity of phobia symptoms, from approaching a few metres from to holding a spider.

SECONDARY OUTCOMES:
Spider Phobia Questionnaire 31 (SPQ-31) | Change from baseline on SPQ-31 (1 week)
  SPQ-31 features 31 spider-focused scenarios which must be answered by a yes/no response, with ascending scores indicative of increased degree of arachnophobia.
Spider Phobia Questionnaire 31 (SPQ-31) | Change from baseline on SPQ-31 (12 week)
  SPQ-31 features 31 spider-focused scenarios which must be answered by a yes/no response, with ascending scores indicative of increased degree of arachnophobia.
Spider Phobia Questionnaire 31 (SPQ-31) | Change from baseline on SPQ-31 (52 week)
  SPQ-31 features 31 spider-focused scenarios which must be answered by a yes/no response, with ascending scores indicative of increased degree of arachnophobia.
Spider Phobia Questionnaire 31 (SPQ-31) | Change from baseline on SPQ-31 (3 year)
  SPQ-31 features 31 spider-focused scenarios which must be answered by a yes/no response, with ascending scores indicative of increased degree of arachnophobia.
Fear of Spiders Questionnaire 18 (FSQ-18) | Change from baseline in FSQ-18 (1 week)
  FSQ-18 features 18 questions about fear and avoidance of spiders.
Fear of Spiders Questionnaire 18 (FSQ-18) | Change from baseline in FSQ-18 (12 week)
  FSQ-18 features 18 questions about fear and avoidance of spiders.
Fear of Spiders Questionnaire 18 (FSQ-18) | Change from baseline in FSQ-18 (52 week)
  FSQ-18 features 18 questions about fear and avoidance of spiders.
Fear of Spiders Questionnaire 18 (FSQ-18) | Change from baseline in FSQ-18 (3 year)
  FSQ-18 features 18 questions about fear and avoidance of spiders.
Generalized Anxiety Disorder Assessment 7 (GAD-7) | Change from baseline in GAD-7 (1 week)
  GAD-7 features seven items for assessing anxiety and screening for generalized anxiety disorder.
Generalized Anxiety Disorder Assessment 7 (GAD-7) | Change from baseline in GAD-7 (12 week)
  GAD-7 features seven items for assessing anxiety and screening for generalized anxiety disorder.
Generalized Anxiety Disorder Assessment 7 (GAD-7) | Change from baseline in GAD-7 (52 week)
  GAD-7 features seven items for assessing anxiety and screening for generalized anxiety disorder.
Generalized Anxiety Disorder Assessment 7 (GAD-7) | Change from baseline in GAD-7 (3 year)
  GAD-7 features seven items for assessing anxiety and screening for generalized anxiety disorder.
Patient Health Questionnaire 9 (PHQ-9) | Change from baseline in PHQ-9 (1 week)
  PHQ-9 features nine items for assessing depression in a clinical context and screening of depression in the general population.
Patient Health Questionnaire 9 (PHQ-9) | Change from baseline in PHQ-9 (12 week)
  PHQ-9 features nine items for assessing depression in a clinical context and screening of depression in the general population.
Patient Health Questionnaire 9 (PHQ-9) | Change from baseline in PHQ-9 (52 week)
  PHQ-9 features nine items for assessing depression in a clinical context and screening of depression in the general population.
Patient Health Questionnaire 9 (PHQ-9) | Change from baseline in PHQ-9 (3 year)
  PHQ-9 features nine items for assessing depression in a clinical context and screening of depression in the general population.
Brunnsviken Brief Quality of Life Scale (BBQ) | Change from baseline in BBQ (1 week)
  BBQ features 12 items concerning 6 areas of life rated on importance and satisfaction.
Brunnsviken Brief Quality of Life Scale (BBQ) | Change from baseline in BBQ (12 week)
  BBQ features 12 items concerning 6 areas of life rated on importance and satisfaction.
Brunnsviken Brief Quality of Life Scale (BBQ) | Change from baseline in BBQ (52 week)
  BBQ features 12 items concerning 6 areas of life rated on importance and satisfaction.
Brunnsviken Brief Quality of Life Scale (BBQ) | Change from baseline in BBQ (3 year)
  BBQ features 12 items concerning 6 areas of life rated on importance and satisfaction.
Diagnostic criteria for specific phobia according to interview (DSM-5) | Change from baseline for specific phobia (DSM-5) (12 weeks)
Diagnostic criteria for specific phobia according to interview (DSM-5) | Change from baseline for specific phobia (DSM-5) (52 weeks)
Diagnostic criteria for specific phobia according to interview (DSM-5) | Change from baseline for specific phobia (DSM-5) (3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, PhD, Principal Investigator — Stockholm University
Locations (1):
- Department of Psychology, Stockholm, Sweden

REFERENCES:
- [Result] Miloff A, Lindner P, Dafgard P, Deak S, Garke M, Hamilton W, Heinsoo J, Kristoffersson G, Rafi J, Sindemark K, Sjolund J, Zenger M, Reuterskiold L, Andersson G, Carlbring P. Automated virtual reality exposure therapy for spider phobia vs. in-vivo one-session treatment: A randomized non-inferiority trial. Behav Res Ther. 2019 Jul;118:130-140. doi: 10.1016/j.brat.2019.04.004. Epub 2019 Apr 16. PMID 31075675
- [Derived] Miloff A, Lindner P, Hamilton W, Reuterskiold L, Andersson G, Carlbring P. Single-session gamified virtual reality exposure therapy for spider phobia vs. traditional exposure therapy: study protocol for a randomized controlled non-inferiority trial. Trials. 2016 Feb 2;17:60. doi: 10.1186/s13063-016-1171-1. PMID 26833396